CLINICAL TRIAL: NCT03105934
Title: Repeatability of Optical Coherence Tomography (OCT) and Intravascular Ultrasound (IV-US) in Pulmonary Arterial Hypertension
Brief Title: Repeatability of OCT and IV-US in Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IVUS
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — hydralazine 4-anisaldehyde hydrazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Arterial Hypertension (Experimental): Patients with Pulmonary Arterial Hypertension
  Interventions: Procedure: Patients with Pulmonary Arterial Hypertension

INTERVENTIONS:
Procedure: Patients with Pulmonary Arterial Hypertension — 2 repeated measurement session to enable assessment of technical and medium-term reproducibility of IV-US and IV-OCT.

SUMMARY:
To assess the correlation between pulmonary IV-OCT and pulmonary IV-US measurements and standard PAH clinical measures of disease progression and the relative sensitivity of the techniques to change.

ELIGIBILITY:
Inclusion Criteria:

* With confirmed diagnosis of PAH Group 1 according to the ESC/ERS Guidelines
* With severe disease, defined as Class II- III of the modified WHO functional classes in the ESC/ERS Guidelines

Exclusion Criteria:

* That according to investigator criteria cannot participate in the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Image measurements | 12 months
  Repeat acquisitions to be made in the same regions and in locations

CONTACTS AND LOCATIONS:
Overall Officials: Enric Domingo, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain